CLINICAL TRIAL: NCT04984837
Title: A Randomized Non Comparative Phase II Study of Lacutamab With GemOx Versus GemOx Alone in Relapsed/Refractory Patients With Peripheral T-cell Lymphoma
Brief Title: Study of Lacutamab in Peripheral T-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KILT
Record Dates: First submitted 2021-07-18; First posted 2021-08-02 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Peripheral T Cell Lymphoma; Relapse/Recurrence
Keywords: KIR3DL2; PTCL; T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Recurrence; Lymphoma, T-Cell | interventions — Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lacutamab (Experimental): Lacutamab 750 mg/IV + GEmOx (1000 mg/m² / 100 mg/m²) 6 cycles of 3 weeks (4,5 months) during the induction phase Lacutamab 750 mg/IV for a maximum of 20 additional cycles of 4 weeks during the maintenance phase
  Interventions: Drug: Lacutamab; Drug: Gemcitabine; Drug: Oxaliplatine
- Standard of care (Active Comparator): GemOx (1000 mg/m² / 100 mg/m²) 6 cycles of 3 weeks (4,5 months) during the induction phase
  Interventions: Drug: Gemcitabine; Drug: Oxaliplatine

INTERVENTIONS:
Drug: Lacutamab — 750 mg/IV
  Arms: Lacutamab
Drug: Gemcitabine — 1000 mg/m²
Drug: Oxaliplatine — 100 mg/m²

SUMMARY:
This is an open-label multicenter randomized non comparative phase II study to evaluate the safety and efficacy of the monoclonal anti-KIR3DL2 antibody Lacutamab in patients with Refractory/Relapsing (R/R) KIR3DL2 positive Peripheral T Cell Lymphoma (PTCL) : Not Other Specified (NOS), PTCL-TFH (including Angioimmunoblastic T-cell Lymphoma (AITL), Follicular T-cell lymphoma, Nodal peripheral T-cell lymphoma with TFH phenotype), Anaplastic large cell lymphoma (ALCL), Adult T-cell leukemia/lymphoma (ATL), Hepatosplenic T-cell lymphoma (HSTL), Enteropathy-associated T-cell lymphoma (EATL), Monomorphic epitheliotropic intestinal T cell lymphoma (MEITL), NK-T cell lymphoma (NKT) and Aggressive NK-cell leukemia (ANKL).

The design is non comparative meaning that non comparison between arms will be performed as the control arm will ensure that the assumptions used for sample size calculation are verified. For that reason, randomization is unbalanced in favor of the experimental arm (2:1).

ELIGIBILITY:
Inclusion Criteria:

* 1. KIR3DL2-positive with at least 1% of tumour cells positivity, before randomization, based on central evaluation by immunohistochemistry (IHC) 2. Patients with histologically documented PTCL:

  * Biopsy-proven treated PTCL defined by the WHO 2016 criteria (the biopsy at relapse is recommended but not mandatory):

    * PTCL-NOS
    * PTCL-TFH (AITL, Follicular T-cell lymphoma, Nodal peripheral T-cell lymphoma with TFH phenotype)
    * ALCL
    * ATL: acute- or lymphoma-type
    * HSTL
    * EATL
    * MEITL
    * NKT
    * ANKL 3. For patients with ALCL: previously treated with brentuximab vedotin 4. Relapsed/refractory PTCL after at least one previous line of systemic based regimen of chemotherapy (no mandatory latency after the previous treatment) 5. With a maximum of 2 prior lines of systemic therapies, including autologous stem cell transplantation (ASCT is authorized in first and second line and is not counted as a unique line, even if associated to a systemic therapy) 6. Bi-dimensionally measurable disease defined by at least one single node or tumor lesion ≥ 1.5 cm assessed by CT scan 7. Signed written screening informed consent prior to KIR3DL2 screening 8. Signed written study informed consent prior to randomization 9. Aged 18 years or more with no upper age limit, at randomization 10. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 3 prior to prephase treatment (if applicable), and 0 to 2 prior randomization 11. Minimum life expectancy of 3 months 12. Females of childbearing potential (FCBP) must agree to use highly effective contraceptive method* from C1D1, during the entire study period, during dose interruptions, and for 9 months after the last study treatments 13. FCBP must have a negative serum or urinary pregnancy test within 28 days prior C1D1 14. Male patients and their partner (FCBP) must agree to use two reliable forms of contraception (condom for males and hormonal method for partners) from C1D1, during the entire study period, during dose interruptions, and for 9 months after the last study treatments

Exclusion Criteria:

* 1. Patients with active COVID-19 infection (last positive PCR < 2 weeks before randomization) 2. Patients taking immunotherapy or chemotherapy, except short-term corticosteroids in monotherapy at a cumulated dose equivalent of prednisone ≤ 1mg/kg/day, during 7 consecutive days, within 3 weeks prior to first administration of study drug (C1D1); or prephase treatment given at investigator's discretion before randomization and for maximum 3 weeks (glucocorticosteroids, vepesid (VP16), cyclophosphamide, vincristine and prednisone (COP)) 3. Previous treatment by Gemcitabine or Oxaliplatin 4. Use of any experimental anti-cancer drug therapy within 6 weeks before randomization 5. Contraindication to any drug contained in the study treatment regimen 6. Previous allogenic hematopoietic cell transplantation 7. Positive test results for HIV and Hepatitis C Virus (HCV) (Patients who are positive for HCV antibody must be negative for HCV by PCR to be eligible for study participation) 8. Known active hepatitis B (positive Ag HBs) (if latent Hepatitis B Virus (HBV) (positive anti-HBc), patients have to be treated with Entecavir (Baraclude ®) and HBV PCR should be performed every month to allow antiviral strategy adaptation) 9. Central nervous system or meningeal involvement by lymphoma 10. Any of the following laboratory abnormalities prior randomization:

  * Absolute neutrophil count (ANC) < 1 G/L, unless neutropenia is related to PTCL
  * Platelet count < 75 G/L, unless thrombopenia is related to PTCL
  * Alkaline Phosphatases > 2.5 x upper limit of normal (ULN)
  * Serum Glutamoyl-oxaloacetate Transferase (SGOT) /Alanine aminotransferase (AST) or Serum Glutamate Pyruvate Transaminase (SGPT)/Alanine aminotransferase (ALT) > 2.5 x ULN
  * Bilirubin > 1.5 x ULN, unless SGOT/AST and SGPT/ALT > 2.5 x ULN or bilirubin elevated due to PTCL or hemolysis
  * Calculated creatinine clearance (MDRD or Cockcroft) < 40 mL/min 11. Any significant cardiovascular impairment: New York Heart Association (NYHA) Class III or IV cardiac disease, uncontrolled high blood pressure, unstable angina, myocardial infarction or stroke within the last 6 months from randomization, and cardiac arrhythmia within the last 3 months from randomization 12. Uncontrolled clinically significant intercurrent illness including, but not limited to, diabetes, ongoing active infections. Patients receiving antibiotics for infections that are under control may be included in the study 13. Concurrent malignancy or prior history of malignancies other than lymphoma unless the subject has been free of disease for ≥ 2 years, except early stage cutaneous squamous or basal cell carcinoma, localized prostate cancer, or cervical intraepithelial neoplasia 14. Major surgery within 4 weeks before randomization 15. Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
median modified progression-free survival (mPFS) - CT-based | 5,5 years.
  time from randomization until one of the following events occurs, whichever comes first:
  1. Disease progression (PD)
  2. Administration of any additional unplanned anti-lymphoma treatment (except allogeneic or autologous hematopoietic cell transplantations (HCT))
  3. Relapse after achievement of CR
  4. Death due to any cause. PD and relapse will be evaluated according to Lugano 2014 criteria (CT-based).

SECONDARY OUTCOMES:
median modified progression-free survival (mPFS) - PET-based | 5,5 years.
Number of Adverse Events | 5,5 years.
overall survival (OS) | 5,5 years.
complete response rate (CRR) Lugano 2014 criteria (CT-based) | 5,5 years.
complete response rate (CRR) Lugano 2014 criteria (PET-based) | 5,5 years.
overall response rate (ORR) Lugano 2014 criteria (CT-based) | 5,5 years.
overall response rate (ORR) Lugano 2014 criteria (PET-based) | 5,5 years.
response rate assessed by Deauville criteria | 5,5 years.
duration of response (DOR), | 5,5 years.
  1. Disease progression (PD)
  2. Administration of any additional unplanned anti-lymphoma treatment (except allogeneic or autologous hematopoietic cell transplantations (HCT))
  3. Relapse after achievement of CR
  4. Death due to any cause
rate of patients proceeding to allogenic stem cell transplantation | 5,5 years.
Pharmacokinetics of lacutamab with GemOx : Maximal Concentration of lacutamab (Cmax) | 1 month (1 cycle)
Pharmacokinetics of lacutamab with GemOx : Trough Concentration of lacutamab (Ctrough) | 1 month (1 cycle)
Pharmacokinetics of lacutamab with GemOx : Maximal Concentration of lacutamab (Cmax) | 2 months (2 cycles)
Pharmacokinetics of lacutamab with GemOx : Trough Concentration of lacutamab (Ctrough) | 2 months (2 cycles)
Pharmacokinetics of lacutamab with GemOx : Maximal Concentration of lacutamab (Cmax) | 3 months (3 cycles)
Pharmacokinetics of lacutamab with GemOx : Trough Concentration of lacutamab (Ctrough) | 3 months (3 cycles)
Pharmacokinetics of lacutamab with GemOx : Maximal Concentration of lacutamab (Cmax) | 7 months (7 cycles)
Pharmacokinetics of lacutamab with GemOx : Trough Concentration of lacutamab (Ctrough) | 7 months (7 cycles)
Pharmacokinetics of lacutamab with GemOx : Maximal Concentration of lacutamab (Cmax) | 9 months (9 cycles)
Pharmacokinetics of lacutamab with GemOx : Trough Concentration of lacutamab (Ctrough) | 9 months (9 cycles)
Pharmacokinetics of lacutamab with GemOx : Maximal Concentration of lacutamab (Cmax) | 15 months (15 cycles)
Pharmacokinetics of lacutamab with GemOx : Trough Concentration of lacutamab (Ctrough) | 15 months (15 cycles)
Pharmacokinetics of lacutamab with GemOx : Maximal Concentration of lacutamab (Cmax) | 26 months (26 cycles)
Pharmacokinetics of lacutamab with GemOx : Trough Concentration of lacutamab (Ctrough) | 26 months (26 cycles)
Pharmacokinetics of lacutamab with GemOx : Maximal Concentration of lacutamab (Cmax) | 29 months (29 cycles)
Pharmacokinetics of lacutamab with GemOx : Trough Concentration of lacutamab (Ctrough) | 29 months (29 cycles)
Immunogenicity : concentration of Anti-Drug Antibodies (ADA)) of lacutamab with GemOx | 1 month (1 cycle)
Immunogenicity : concentration of Anti-Drug Antibodies (ADA)) of lacutamab with GemOx | 2 months (2 cycles)
Immunogenicity : concentration of Anti-Drug Antibodies (ADA)) of lacutamab with GemOx | 3 months (3 cycles)
Immunogenicity : concentration of Anti-Drug Antibodies (ADA)) of lacutamab with GemOx | 7 months (7 cycles)
Immunogenicity : concentration of Anti-Drug Antibodies (ADA)) of lacutamab with GemOx | 9 months (9 cycles)
Immunogenicity : concentration of Anti-Drug Antibodies (ADA)) of lacutamab with GemOx | 15 months (15 cycles)
Immunogenicity : concentration of Anti-Drug Antibodies (ADA)) of lacutamab with GemOx | 26 months
Immunogenicity : concentration of Anti-Drug Antibodies (ADA)) of lacutamab with GemOx | 29 months

CONTACTS AND LOCATIONS:
Overall Officials: Morgane Cheminant, Study Chair — Lymphoma Study Association
Locations (64):
- Belgium (12):
  - Institut Jules Bordet, Anderlecht
  - VZW ZAS, Antwerp
  - A. Z. Sint-Jan, Bruges
  - Cliniques Universitaires de Bruxelles - Hôpital Erasme, Brussels
  - Cliniques universitaires Saint-Luc - Université catholique de Louvain, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - UZ Antwerpen, Edegem
  - HELORA - Hôpital de La LouvièreSite Jolimont, Haine-Saint-Paul
  - CHU de LIEGE - Domaine Sart Tilman, Liège
  - Clinique CHC MontLégia, Liège
  - CHR Verviers, Verviers
  - CHU Dinant Godinne - UCL Namur - YVOIR, Yvoir
- France (43):
  - CHU de Nancy - Brabois, Nancy, France
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - CH d Avignon - Hopital Henri Duffaut, Avignon
  - CH de la Côte Basque - Hôpital de Bayonne, Bayonne
  - Institut Bergonié, Bordeaux
  - CHU de Caen - Côte de Nacre - IHBN, Caen
  - CH Métropole Savoie, Chambéry
  - CHU de Clermont Ferrand - Estaing, Clermont-Ferrand
  - APHP - Hôpital Henri Mondor, Créteil
  - CHU de Dijon BOURGOGNE - Hôpital François Mitterand, Dijon
  - CH de Dunkerque, Dunkirk
  - CHD de Vendée, La Roche-sur-Yon
  - CHU de Grenoble - Hôpital Albert Michallon, La Tronche
  - Ch de Versailles - Hopital Andre Mignot, Le Chesnay
  - CH du Mans, Le Mans
  - CHRU de Lille - Hôpital Claude Hurriez, Lille
  - Hôpital Saint Vincent-De-Paul, Lille
  - Chu de Limoges - Hopital Dupuytren, Limoges
  - Centre Leon Berard, Lyon
  - Chu de Meaux, Meaux
  - CHU de Montpellier, Montpellier
  - CH de Mulhouse, Mulhouse
  - CHU de Nantes - Hôtel Dieu, Nantes
  - CHU de Nîmes, Nîmes
  - CHR d'Orléans, Orléans
  - APHP - Hopital Necker, Paris
  - APHP - Hôpital de la Pitié Salpétrière, Paris
  - APHP - Hôpital Saint Antoine, Paris
  - APHP - Hôpital Saint Louis, Paris
  - CH de Perpignan, Perpignan
  - CHU de Bordeaux - Hôpital Haut Lévêque - Centre François Magendie, Pessac
  - CH de Périgueux, Périgueux
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Poitiers - Hôpital de La Milétrie, Poitiers
  - Centre Hospitalier Annecy Genevois, Pringy
  - CHU de Reims, Reims
  - CHU de Rennes - Hôpital de Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie et d'Hématologie Universitaire de Saint-Étienne, Saint-Etienne
  - Institut de Cancerologie Strasbourg Europe, Strasbourg
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse
  - CH de Bretagne Atlantique - Hopital Chubert, Vannes
- Germany (5):
  - Charite Universitat Smedizin Berlin, Berlin
  - GEORG-AUGUST-UNIV, GOETTINGEN - Klinik fur Haematologie und Medizini, Goettigen
  - Universitatsklinikum Halle (Saale), Halle
  - UNIVERSITAT LEIPZIG - Klinik fur Hamatologie, Zelltherapie und Hamostaseo, Leipzig
  - UNIVERSITATSKLINIKUM REGENSBURG - Klinik für Innere Medizin III, Regensburg
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz - Hematologia, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheminant M, Lhermitte L, Bruneau J, Sicard H, Bonnafous C, Touzart A, Bourbon E, Ortonne N, Genestier L, Gaulard P, Palmic P, Suarez F, Frenzel L, Naveau L, Bazarbachi A, Dussiot M, Waast L, Avettand-Fenoel V, Brouzes C, Pique C, Lepelletier Y, Asnafi V, Marcais A, Hermine O. KIR3DL2 contributes to the typing of acute adult T-cell leukemia and is a potential therapeutic target. Blood. 2022 Sep 29;140(13):1522-1532. doi: 10.1182/blood.2022016765. PMID 35687761